CLINICAL TRIAL: NCT02945553
Title: Prevention of Skeletal Muscle Adaptations to Traumatic Knee Injury and Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Michael J. Toth, Ph.D., Associate Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: M16-609
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-11

CONDITIONS: Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NMES (Experimental): Neuromuscular electrical stimulation (NMES) group
  Interventions: Device: Neuromuscular electrical stimulation
- Microstimulation (Active Comparator): Microstimulation
  Interventions: Device: Microstimulation

INTERVENTIONS:
Device: Neuromuscular electrical stimulation — Neuromuscular electrical stimulation (NMES) will be performed 5 times/week for one hour each day. NMES will start within 1 week of injury and continue till 3 weeks following surgery.
  Arms: NMES
Device: Microstimulation — Microstimulation will be performed 5 times/week for one hour each day. Microstimulation will start within 1 week of injury and continue till 3 weeks following surgery.
  Arms: Microstimulation

SUMMARY:
Traumatic knee injury is common and highly debilitating. Surgical reconstruction/repair improves knee biomechanics and function, but neuromuscular dysfunction persist for years despite rehabilitation, hindering resumption of normal activities, increasing risk of further injury and, in a majority of patients, hastening the development of knee osteoarthritis (OA). Our goal in this research study is to evaluate the utility of neuromuscular electrical stimulation (NMES), initiated following injury and maintained through the early post-surgical period, to prevent muscle atrophy and intrinsic contractile dysfunction compared to active control intervention of micro-electrical stimulation.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 yrs
* BMI <35 kg/m2
* acute, first-time, ACL rupture with or without meniscus injury
* scheduled to undergo reconstruction with a BPTB autograft

Exclusion Criteria:

* history of prior knee/lower extremity surgery or non-surgical intervention (eg, intra-articular injection) on either leg
* abnormal laxity of any lower extremity ligament other than the injured ACL
* signs or symptoms of arthritis, autoimmune or inflammatory disease or diabetes
* grade IIIb or greater articular cartilage lesions (ICRS criteria)
* women who are/plan on becoming pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Toth, Ph.D., Principal Investigator — University of Vermont; Bruce D. Beynnon, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- University of Vermont College of Medicine, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Yes
Research data (deidentified) which documents, supports and validates research findings will be stored on the University of Vermont College of Medicine computer system and will be made available upon final acceptance for publication of the major findings from the proposed studies. This includes raw data generated from all clinical and laboratory-based assessments under a data-sharing agreement.

REFERENCES:
- [Derived] Toth MJ, Tourville TW, Voigt TB, Choquette RH, Anair BM, Falcone MJ, Failla MJ, Stevens-Lapslaey JE, Endres NK, Slauterbeck JR, Beynnon BD. Utility of Neuromuscular Electrical Stimulation to Preserve Quadriceps Muscle Fiber Size and Contractility After Anterior Cruciate Ligament Injuries and Reconstruction: A Randomized, Sham-Controlled, Blinded Trial. Am J Sports Med. 2020 Aug;48(10):2429-2437. doi: 10.1177/0363546520933622. Epub 2020 Jul 6. PMID 32631074

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment started in October 2016 and ended in December 2018. Patients were enrolled from an academic orthopedic surgical clinic.
Period: Overall Study
Arm/Group | NMES | Microstimulation
Started | 14 | 11
Completed | 11 (Included in analysis for primary aim.) | 9 (Included in analysis for primary aim.)
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Population: Three (3) patients in NMES and two (2) patients in microstimulation groups were lost to follow-up for analyses of primary aim.
Groups:
- Total: Total of all reporting groups
Arm/Group | NMES | Microstimulation | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 25
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 11 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 10 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 11 | 25
Type of Injury [Count of Participants; unit: Participants]
  ACL rupture only | 3 | 4 | 7
  ACL rupture + Meniscus injury | 3 | 1 | 4
  ACL rupture + Meniscus injury + Cartilage injury | 4 | 1 | 5
  Exclusion found at surgery (Avulsion) | 1 | 1 | 2
  Withdrew prior to surgery | 1 | 1 | 2
  ACL rupture + Cartilage | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Cross-sectional Area of Skeletal Muscle Fibers (All Fibers)
Description: Cross-sectional area of skeletal muscle fibers will be evaluated using immunohistochemistry, with specification of all relevant muscle fiber types
Time Frame: Difference between injured and non-injured leg at 3 weeks post-surgery
Measure: Mean (Standard Error); unit: micrometer squared
Arm/Group | NMES | Microstimulation
Number analyzed (Participants) | 11 | 9
micrometer squared
  Non-injured leg | 2827 (141) | 3318 (153)
  Injured leg | 2206 (125) | 2376 (130)
Statistical Analysis 1: Comparison: NMES vs Microstimulation; Test type: Other — Mixed model analysis of variance; p < 0.05, ANOVA; Mean Difference (Final Values) = 1596, Standard Deviation 202

2. Primary Outcome: Maximal Calcium-activated Tension Single Muscle Fiber Tension (Myosin Heavy Chain (MHC) IIA Fibers)
Description: Tension (force per unit muscle fiber cross-sectional area) from segments of chemically-skinned single human muscle fibers will be assessed under maximal calcium-activated condition, with muscle fiber type determined post-measurement by gel electrophoresis
Time Frame: Difference between injured and non-injured leg at 3 weeks post-surgery
Population: Difference in sample size in NMES group is due to the fact that one volunteer did not have sufficient tissue to allow assessment of muscle fiber mechanical properties.
Measure: Mean (Standard Error); unit: mN/mm2
Arm/Group | NMES | Microstimulation
Number analyzed (Participants) | 10 | 9
mN/mm2
  Injured leg | 127 (7) | 137 (8)
  Non-injured leg | 169 (7) | 175 (7)

3. Primary Outcome: Maximal Single Muscle Fiber Shortening Velocity (Myosin Heavy Chain (MHC) IIA Fibers)
Description: Maximal shortening velocity from segments of chemically-skinned single human muscle fibers will be assessed, with muscle fiber type determined post-measurement by gel electrophoresis
Time Frame: Difference between injured and non-injured leg at 3 weeks post-surgery
Population: as for outcome 2
Measure: Mean (Standard Error); unit: muscle length per second (ML/s)
Groups:
- Microstimulation: Sham control group
- Neuromuscular Electrical Stimlulation: Treatment group
Arm/Group | Microstimulation | Neuromuscular Electrical Stimlulation
Number analyzed (Participants) | 9 | 10
muscle length per second (ML/s)
  Injured leg | 1.74 (0.1) | 1.67 (0.09)
  Non-injured leg | 1.95 (.09) | 1.92 (0.09)

4. Primary Outcome: Cross-sectional Area of Skeletal Muscle Fibers (Myosin Heavy Chain (MHC) I Fibers)
Description: as for outcome 1
Time Frame: Difference between injured and non-injured leg at 3 weeks post-surgery
Measure: Mean (Standard Error); unit: micrometer squared
Groups:
- Microstimulation: Microstimulation: Sham control group
- Neuromuscular Electrical Stimlulation: Neuromuscular electrical stimulation: Treatment group
Arm/Group | Microstimulation | Neuromuscular Electrical Stimlulation
Number analyzed (Participants) | 9 | 11
micrometer squared
  Injured leg | 2552 (134) | 2206 (125)
  Non-injured leg | 3217 (151) | 2827 (141)

5. Primary Outcome: Cross-sectional Area of Skeletal Muscle Fibers (MHC IIA)
Description: as for outcome 1
Time Frame: Difference between injured and non-injured leg at 3 weeks post-surgery
Measure: Mean (Standard Error); unit: micrometer squared
Arm/Group | Microstimulation | Neuromuscular Electrical Stimlulation
Number analyzed (Participants) | 9 | 11
micrometer squared
  Injured leg | 2290 (170) | 2206 (167)
  Non-injured leg | 3739 (217) | 3318 (204)

6. Secondary Outcome: Knee Extensor Peak Isokinetic Torque
Description: Peak isokinetic torque is measures in injured and non-injurd leg at 60 deg/s using dynamometry
Time Frame: Difference between injured and non-injured leg at 6 months post-surgery
Population: Difference in number of volunteers in analysis is due to loss of patients during 6-month follow-up.
Measure: Mean (Standard Error); unit: % (injured to non-injured leg)
Arm/Group | Microstimulation | Neuromuscular Electrical Stimlulation
Number analyzed (Participants) | 7 | 9
% (injured to non-injured leg) | 59.4 (7.5) | 66.4 (6.5)
Statistical Analysis 1: Comparison: Microstimulation vs Neuromuscular Electrical Stimlulation; Test type: Other; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 30

ADVERSE EVENTS:
Time Frame: 6 months post-surgery
Description: Adverse event - any untoward or unfavorable medical occurrence, including any abnormal sign (e.g. abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participants' involvement in the research, whether or not considered related to participation in the research.
Arm/Group | Microstimulation | Neuromuscular Electrical Stimlulation
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/14
Other Adverse Events (participants affected / at risk) | 2/11 | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microstimulation (N=11) | Neuromuscular Electrical Stimlulation (N=14)
Re-injury of ACL (graft failure) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient re-injured ACL/tore ACL graft several weeks after completing final study assessments while engaging in sporting activity.
Re-injury of meniscus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient re-injured damaged meniscus during 6-month post-surgery follow-up.
Muscle strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Patient experienced muscle strain during muscle strength assessment.
Procedural complication. (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Patient developed rash related to antiseptic used during muscle biopsy procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT02945553/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT02945553/SAP_001.pdf